CLINICAL TRIAL: NCT07152171
Title: Pain Neuroscience Education Delivered During Aerobic Exercise Versus Exercise Alone in Chronic Low Back Pain
Brief Title: Pain Neuroscience Education Delivered During Aerobic Exercise Versus Exercise Alone
Acronym: PNE-MOVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, RODRIGO NUNEZ, Assistant Professor, PhD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0469
Record Dates: First submitted 2025-08-21; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low Back Pain
Keywords: Musculoskeletal Pain; Pain Neuroscience Education; Aerobic Exercise; Physical Therapy; Rehabilitation
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a two-arm, single-center randomized controlled trial with parallel assignment. Participants with chronic low back pain will be randomized (1:1) to receive either pain neuroscience education delivered during aerobic cycling exercise or aerobic exercise alone. Outcome assessors will be blinded to group allocation.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group allocation. Participants and care providers cannot be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education During Aerobic Exercise (Experimental): Participants will perform 20-30 minutes of supervised aerobic exercise on a cycle ergometer at light intensity (Borg CR10 = 3; 40-50% HRmax). During cycling, they will receive interactive pain neuroscience education covering neurobiology of pain, central sensitization, and self-management strategies. Education will be delivered by a therapist using metaphors and visual aids to facilitate understanding while exercising.
  Interventions: Behavioral: Pain Neuroscience Education During Aerobic Exercise
- Aerobic Exercise Alone (Active Comparator): Participants will perform 20-30 minutes of supervised aerobic exercise on a cycle ergometer at light intensity (Borg CR10 = 3; 40-50% HRmax). No educational content will be provided. Sessions include warm-up, main cycling phase, and cool-down. Exercise parameters (cadence, resistance, and effort perception) will be matched to the experimental group.
  Interventions: Behavioral: Aerobic Exercise Alone

INTERVENTIONS:
Behavioral: Pain Neuroscience Education During Aerobic Exercise — Participants will cycle on an ergometer for 20-30 minutes at light intensity (Borg CR10 = 3; 40-50% HRmax). During cycling, they will receive interactive pain neuroscience education delivered by a therapist, including neurobiology of pain, central sensitization, and self-management strategies. Visual aids and metaphors will be used to facilitate understanding.
  Arms: Pain Neuroscience Education During Aerobic Exercise
Behavioral: Aerobic Exercise Alone — Participants will perform 20-30 minutes of supervised cycling on an ergometer at light intensity (Borg CR10 = 3; 40-50% HRmax). No educational content will be provided. Sessions will include warm-up, main phase, and cool-down, matched in duration and intensity to the experimental group.
  Arms: Aerobic Exercise Alone

SUMMARY:
Chronic musculoskeletal pain is a common health condition that reduces quality of life and increases disability. Pain neuroscience education (PNE) has shown positive effects on pain perception, beliefs, and function, especially when combined with physical activity. This randomized controlled trial will compare the effectiveness of delivering PNE during aerobic exercise on a cycle ergometer versus aerobic exercise alone in patients with chronic musculoskeletal pain.

Participants will be randomly assigned to one of two groups:

PNE during aerobic exercise (experimental group),

Aerobic exercise alone (control group).

Both groups will perform supervised cycling sessions lasting 20-30 minutes at light intensity (Borg CR10 = 3, 40-50% HRmax). The experimental group will simultaneously receive interactive education about pain mechanisms, central sensitization, and self-management strategies, supported by visual aids and metaphors delivered by a therapist during cycling.

Outcomes will be measured at baseline and after the intervention, including:

Pain intensity (Visual Analog Scale),

Pressure pain threshold (algometry),

Functional performance (Sit-to-Stand test),

Perceived effort (Borg CR10),

Safety and comfort (Likert scale),

Muscle activity (surface EMG).

The study will enroll 28 participants (14 per group). The findings are expected to clarify whether integrating education with exercise provides superior benefits compared to exercise alone, offering an innovative, safe, and cost-effective strategy for managing chronic musculoskeletal pain.

DETAILED DESCRIPTION:
Objective To determine whether PNE delivered during cycling exercise produces greater improvements in pain intensity, pain thresholds, and functional outcomes than aerobic exercise alone.

Study Design This is a single-center, randomized controlled trial with two parallel arms (1:1 allocation). A total of 28 participants with chronic musculoskeletal pain will be recruited from the Hospital Clínico de la Universidad de Chile. Randomization will assign 14 participants to the experimental group and 14 to the control group, using the Randomization software (www.randomization.com). The random sequence will be determined prior to the start of the initial assessments and will only be known to an external research assistant with no access to participant characteristics. The assignment will remain hidden and stored in the cloud until the end of the intervention and the collection of all study data. When a participant enrolls in the study, the external research assistant will inform the therapist of the assigned intervention group.

Intervention Experimental group (PNE + exercise): 20-30 minutes of supervised cycling at light intensity (Perceived exertion, Borg CR10 = 3) while receiving interactive PNE. Education covers neurobiology of pain, central sensitization, and self-management, supported by visual aids and metaphors.

Control group (exercise alone): 20-30 minutes of supervised cycling at the same intensity (Perceived exertion, Borg CR10 = 3), without educational content.

Sample Size and Analysis Based on prior effect sizes, 28 participants (14 per group) provide sufficient power to detect moderate differences. Data will be analyzed with mixed-model ANOVA (time × group) and additional parametric or nonparametric tests as appropriate. Statistical significance is set at p < 0.05.

Ethical Considerations The study is approved by the Ethics Committee of Hospital Clínico de la Universidad de Chile. Participants will provide informed consent before participation. Risks are minimal (fatigue or mild discomfort), while expected benefits include improved pain understanding, reduced pain intensity, and improved function. This study will be conducted in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Diagnosis of chronic low back pain lasting ≥ 12 weeks.
* Baseline pain intensity ≥ 4/10 on the Visual Analog Scale (VAS).
* Able to perform light to moderate aerobic exercise
* Willing and able to provide informed consent.

Exclusion Criteria:

* Inability to understand or follow instructions.
* Pregnancy.
* Active cancer diagnosis.
* Neurological disorders affecting the central nervous system (e.g., stroke).
* Participation in alternative or concurrent therapies for pain management.
* History of major orthopedic trauma or surgery in the last 12 months.
* Any medical contraindication to light exercise identified during the medical screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-11-25 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity (Visual Analog Scale, 0-10) | Baseline (pre-session) and immediately post-intervention (within 30 minutes)
  Pain intensity will be assessed using a 10-cm Visual Analog Scale (VAS; 0 = no pain, 10 = worst imaginable pain). The primary endpoint is the change score (post-session minus baseline). Higher scores indicate greater pain.

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold (kgf) by Algometry | Pressure pain threshold (PPT) will be measured at the most symptomatic lumbar region using a handheld algometer. Pressure is increased at a constant rate until the participant first perceives pain; the value (kgf) is recorded. The outcome is the change s
  Baseline (pre-session) and immediately post-intervention (within 30 minutes)
Change in Functional Performance (30-Second Sit-to-Stand Test) | Participants sit on a standard chair (≈43 cm height) with arms crossed and stand up/sit down as many times as possible in 30 seconds. The total number of full stands is recorded. The outcome is the change in repetitions from baseline.
  Baseline (pre-session) and immediately post-intervention (within 30 minutes)
Safety and Comfort Ratings (Likert Scales) | Immediately post-intervention (within 30 minutes)
  Participants rate statements such as "I felt physically comfortable during the session" and "The environment felt safe to exercise" on 5-point Likert scales. Higher scores reflect greater perceived safety/comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No